CLINICAL TRIAL: NCT00985504
Title: A Phase 4, 8-week, Double-blind, Randomized Study Comparing Switching to Duloxetine or Escitalopram in Patients With Major Depressive Disorder and Residual Apathy in the Absence of Depressed Mood
Brief Title: A Study of Patients With Major Depressive Disorder and Residual Apathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13018; F1J-CR-HMGM (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Apathy; Duloxetine Hydrochloride; SSRI; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major; Lethargy | interventions — Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Duloxetine — 60-120 milligrams (mg) taken once daily (QD) by mouth (po) for 8 weeks; with option for additional 2 weeks.
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Escitalopram — 10-20 mg taken QD po for 8 weeks; with option for additional 2 weeks.
  Arms: Escitalopram

SUMMARY:
The purpose of this study is to provide a comparison of the apathy, depression, and functional outcomes associated with switching to duloxetine or escitalopram in patients who have previously responded to treatment with a selective serotonin reuptake inhibitor (SSRI) for major depressive disorder and who have residual apathy in the absence of depressed mood.

DETAILED DESCRIPTION:
Apathy is reported by up to 30% of patients with major depressive disorder (MDD) and is hypothesized to be a treatment emergent adverse effect associated with selective serotonin reuptake inhibitor medication. While there is currently no consistent method for treating apathy among psychiatrists, it has been proposed that switching MDD patients to antidepressant medications containing both serotonin and norepinephrine, such as duloxetine, may reduce the incidence and severity of apathy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Have received treatment with an SSRI (escitalopram, sertraline, paroxetine, or citalopram) for major depressive disorder
* Females of child-bearing potential to test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control
* Apathy Evaluation Scale - Clinician Rated Version (AES-C) total score >30 at screening and randomization.
* Montgomery-Asberg Depression Rating Scale (MADRS) total score ≤15 and Item 1 (apparent sadness) score of <2 at screening and randomization.
* Have a level of understanding sufficient to provide informed consent and to communicate with the investigators, study coordinator, and site personnel.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device
* Have previously completed or withdrawn from this study or any other study investigating duloxetine.
* Have had previous lack of response to an adequate trial of duloxetine within the past 12 months or escitalopram at any time.
* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), diagnosis of mania, bipolar disorder, treatment resistant depression or psychosis; or current suicide risk
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision(DSM-IV-TR),substance abuse or dependence within the 6 months
* Presence of an Axis II disorder
* Monoamine oxidase inhibitor (MAOI) treatment within 14 days prior to randomization or the potential need to use an MAOI during the study
* Positive urine drug screen for any substance of abuse or excluded medication.
* Are pregnant or breast-feeding.
* Serious medical illness, requires hospitalization during the study
* Have uncontrolled narrow-angle glaucoma.
* Have acute liver injury or severe cirrhosis
* Abnormal thyroid stimulating hormone (TSH) concentration
* Amphetamines, dopaminergic medications or modafinil within 14 days prior to randomization or potential need to use such medications during the study or within 14 days of discontinuation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Hill, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glenside, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dandenong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prahran, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba, Canada
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frac. Hacienda de Las Cruces
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douliu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Acute treatment period (1 week): Participants randomized to switch to 60 milligrams (mg) duloxetine once daily (QD) by mouth (po) or 10 mg escitalopram QD po.
  Optimization period (7 weeks): Participants given duloxetine or escitalopram in acute study period may optimize their QD po doses (60-120 mg duloxetine QD po; 10-20 mg escitalopram QD po).
Groups:
- Duloxetine: Participants received 60 milligrams (mg) of duloxetine once daily (QD) by mouth (po) for 1 week (Acute Treatment Period) followed by 60-120 mg QD po for the remaining 7 weeks (Optimization Period), with an option to continue treatment for an additional 2 weeks.
- Escitalopram: Participants received 10 mg of escitalopram QD po for 1 week (Acute Treatment Period) followed by 10-20 mg QD po for the remaining 7 weeks (Optimization Period), with an option to continue treatment for an additional 2 weeks.
Period: Acute Treatment Period
Arm/Group | Duloxetine | Escitalopram
Started | 244 | 239
Completed | 229 | 227
Not Completed | 15 | 12
Not completed — Adverse Event | 3 | 4
Not completed — Entry Criteria Not Met | 1 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Sponsor Decision | 0 | 1
Not completed — Withdrawal by Subject | 9 | 5
Period: Optimization Period
Arm/Group | Duloxetine | Escitalopram
Started | 229 | 227
Completed | 203 | 204
Not Completed | 26 | 23
Not completed — Adverse Event | 7 | 9
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Escitalopram | Total
Number analyzed (Participants) | 244 | 239 | 483
Age Continuous [Mean (Standard Deviation); unit: years] | 44.15 (13.81) | 44.93 (12.89) | 44.54 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 179 | 366
  Male | 57 | 60 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 44 | 89
  Not Hispanic or Latino | 199 | 195 | 394
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants] — One participant selected 2 races. Therefore, the total number of participants in the race category will be larger than the number of participants in the baseline table.
  participants
    American Indian or Alaska Native | 34 | 37 | 71
    Asian | 90 | 82 | 172
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 0 | 1 | 1
    White | 120 | 119 | 239
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 24 | 25 | 49
  Canada | 44 | 43 | 87
  China | 47 | 41 | 88
  Italy | 23 | 22 | 45
  Korea, Republic of | 18 | 15 | 33
  Mexico | 42 | 43 | 85
  Russian Federation | 23 | 25 | 48
  Taiwan | 23 | 25 | 48
Taking Escitalopram 3 Months Prior to Study Entry [Number; unit: participants] — Previous therapy status is defined as the number of participants who had taken escitalopram 3 months prior to study entry.
  participants
    Yes | 67 | 59 | 126
    No | 177 | 180 | 357
Apathy Evaluation Scale - Clinician Rated Version (AES-C) Total Score [Mean (Standard Deviation); unit: units on a scale] — The AES-C is a validated 18-item instrument used to assess cognitive, behavioral, emotional and other symptoms of apathy. Clinicians rate each item based on verbal and nonverbal information provided by the participant. Item scores range from 1 (not at all characteristic) to 4 (a lot characteristic). Total scores range from 18 to 72 where higher derived scores indicate more severe apathy.
  units on a scale | 46.28 (7.82) | 46.34 (8.14) | 46.31 (7.97)
Montgomery-Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  units on a scale | 10.57 (3.49) | 10.29 (3.68) | 10.43 (3.59)
Montgomery-Asberg Depression Rating Scale (MADRS) Item 8 Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS Item 8 assesses participants' inability to feel, through evaluation of their interest in their surroundings or activities that normally give pleasure, as well as their ability to react with adequate emotion to circumstances or people. The score ranges from 0 (normal interest in the surroundings and in other people) to 6 (the experience of being emotionally paralyzed, inability to feel anger, grief or pleasure and a complete or even painful failure to feel for close relatives and friends).
  units on a scale | 1.82 (1.10) | 1.82 (1.15) | 1.82 (1.13)
Clinical Global Impressions of Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
  units on a scale | 3.05 (0.91) | 3.04 (0.91) | 3.05 (0.91)
Rothschild Scale for Antidepressant Tachyphylaxis (RSAT) Total Score [Mean (Standard Deviation); unit: units on a scale] — RSAT assesses symptoms of apathy or decreased motivation among depressed participants who have achieved symptomatic remission with antidepressant treatment and consists of 6 self-report items assessing energy level, motivation and interest, cognitive functioning, weight gain, sleep and sexual functioning, as well as affect. Each item score ranges from 0 to 4 with total scores ranging from 0 to 28. Higher scores indicate greater disease severity.
  units on a scale | 10.72 (4.92) | 10.51 (4.95) | 10.62 (4.93)
The Massachusetts General Hospital Cognitive and Physical functioning Questionnaire (MGH-CPFQ) Total [Mean (Standard Deviation); unit: units on a scale] — The MGH-CPFQ is a 7-item participant-rated questionnaire evaluating the participant's cognitive and physical well-being during the past month. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each of the 7 items is scored on a 6-point scale ranging from "greater than normal" (score of 1) to "normal" (score of 2), to "totally absent" (score of 6). Total scores range from 7 to 42. Higher scores indicate greater disease severity.
  units on a scale | 24.78 (5.73) | 24.69 (5.83) | 24.73 (5.78)
Sheehan Disability Scale - Total Score (SDS Total) [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
  units on a scale | 15.32 (6.76) | 14.62 (6.39) | 14.98 (6.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Apathy Evaluation Scale - Clinician Rated Version (AES-C) Total Score at Week 8
Description: The AES-C is a validated 18-item instrument used to assess cognitive, behavioral, emotional and other symptoms of apathy. Clinicians rate each item based on verbal and nonverbal information provided by the participant. Item scores range from 1 (not at all characteristic) to 4 (a lot characteristic). Total scores range from 18 to 72 where higher derived scores indicate more severe apathy. The Least Squares (LS) Mean Value was calculated from a mixed model repeated measures (MMRM) model with terms of treatment, pooled investigator, visit, treatment*visit, baseline, and baseline*visit.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 213 | 210
units on a scale | -13.88 (0.54) | -13.50 (0.54)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.612, Mixed Models Analysis; The "Kenward-Roger approximation" was used in the MMRM model; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.87 to 1.10]

2. Secondary Outcome: Change From Baseline in the Apathy Evaluation Scale-Clinician Rated Version (AES-C) Subscale Scores at Week 8
Description: AES-C subscales separately assess participants' intensity of cognitive, behavioral, emotional, and other apathy symptoms with individual item scores of 1 (not at all characteristic) to 4 (a lot characteristic). Subtotal score ranges for the subscales are: 8-32 (cognitive), 5-20 (behavioral), 2-8 (emotional), and 3-12 for other (display of personal insight, initiative and motivation). Higher subscale scores indicate greater illness severity. The LS Mean Value was calculated from an MMRM model with terms of treatment, pooled investigator, visit, treatment*visit, baseline, and baseline*visit.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 213 | 210
units on a scale
  Cognition Items Total Score | -6.49 (0.26) | -6.25 (0.26)
  Behavior Items Total Score | -3.35 (0.15) | -3.25 (0.16)
  Emotional Items Total Score | -1.66 (0.08) | -1.58 (0.08)
  Other Items Total Score | -2.43 (0.10) | -2.44 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.504, Mixed Models Analysis — This is the p-value for Cognition Items Total Score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 2: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.665, Mixed Models Analysis — This is the p-value for the Behavior Items Total Score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 3: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.489, Mixed Models Analysis — This is the p-value for Emotional Items Total Score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 4: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.945, Mixed Models Analysis — This is the p-value for Other Items Total Score; The "Kenward-Roger approximation" was used in the MMRM model

3. Secondary Outcome: Change From Baseline in the Rothschild Scale for Antidepressant Tachyphylaxis (RSAT) Total and Individual Item Scores at Week 8
Description: RSAT assesses symptoms of apathy or decreased motivation among depressed participants who have achieved symptomatic remission with antidepressant treatment and consists of 6 self-report items assessing energy level, motivation and interest, cognitive functioning, weight gain, sleep and sexual functioning, as well as affect. Each item score ranges from 0 to 4 with total scores ranging from 0 to 28. Higher scores indicate greater disease severity. LS Mean Value was calculated from an MMRM model with terms of treatment, pooled investigator, visit, treatment*visit, baseline, and baseline*visit.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline at and least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 212 | 210
units on a scale
  RSAT Total Score | -5.50 (0.26) | -4.98 (0.26)
  Energy Level | -1.33 (0.07) | -1.19 (0.07)
  Motivation and Interest | -1.41 (0.06) | -1.29 (0.06)
  Cognitive Functioning | -0.90 (0.06) | -0.80 (0.06)
  Weight Gain | -0.25 (0.05) | -0.11 (0.05)
  Sleep | -0.48 (0.08) | -0.55 (0.08)
  Sexual Functioning | -0.62 (0.07) | -0.60 (0.07)
  Affect | -0.53 (0.04) | -0.50 (0.04)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.157, Mixed Models Analysis — This is the p-value for the Total Score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 2: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.119, Mixed Models Analysis — This is the p-value for the Energy Level score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 3: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.184, Mixed Models Analysis — This is the p-value for the Motivation and Interest score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 4: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.226, Mixed Models Analysis — This is the p-value for the Cognitive Functioning score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 5: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — This is the p-value for the Weight Gain score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 6: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.466, Mixed Models Analysis — This is the p-value for the Sleep score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 7: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis — This is the p-value for the Sexual Functioning score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 8: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.599, Mixed Models Analysis — This is the p-value for the Affect score; The "Kenward-Roger approximation" was used in the MMRM model

4. Secondary Outcome: Patient's Global Impressions of Improvement Scale (PGI-I) Rating Scale Score at Week 8
Description: The PGI-I is a scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). The LS Mean Value was calculated from an MMRM model with terms of treatment, pooled investigator, visit, and treatment*visit.
Time Frame: 8 weeks
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 213 | 210
units on a scale | 2.59 (0.08) | 2.55 (0.08)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — This is the p-value for the PGI-I; The "Kenward-Roger approximation" was used in the MMRM model

5. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity (CGI-S) Rating Scale at Week 8
Description: The CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The LS Mean Value was calculated from an MMRM model with terms of treatment, pooled investigator, visit, treatment*visit, baseline, and baseline*visit.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 213 | 210
units on a scale | -0.86 (0.06) | -0.93 (0.06)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.410, Mixed Models Analysis; The "Kenward-Roger approximation" was used in the MMRM model

6. Secondary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Item 8 (Inability to Feel) at Week 8
Description: MADRS is a rating scale for severity of depressive mood symptoms and has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Item 8 assesses the participant's inability to feel. Scores range from 0 (normal interest in surroundings and other people) to 6 (emotional paralysis, inability to feel anger/grief/pleasure). The LS Mean Value was calculated from an MMRM model with terms of treatment, pooled investigator, visit, treatment*visit, baseline, and baseline*visit.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 213 | 210
units on a scale
  Total Score | -4.21 (0.32) | -4.14 (0.33)
  Item 8 (Inability to Feel) | -1.01 (0.06) | -0.90 (0.06)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.880, Mixed Models Analysis — This is the p-value for the Total Score; The "Kenward-Roger approximation" was used in the MMRM model
Statistical Analysis 2: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.224, Mixed Models Analysis — This is the p-value for the Item 8 (Inability to Feel) score; The "Kenward-Roger approximation" was used in the MMRM model

7. Secondary Outcome: Change From Baseline in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) Total and Item Scores at Week 8
Description: The MGH-CPFQ is a 7-item participant-rated questionnaire evaluating the participant's cognitive and physical well-being during the past month. The MGH-CPFQ assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item is scored on a 6-point scale ranging from 1 ("greater than normal") to 2 ("normal") to 6 ("totally absent"). Total scores range from 7 to 42. Higher scores indicate greater disease severity. The LS Mean Value was calculated from an analysis of covariance (ANCOVA) model with terms of treatment, pooled investigator, and baseline.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 221 | 214
units on a scale
  Total Score | -6.96 (0.34) | -6.91 (0.35)
  Motivation/Interest/Enthusiasm Score | -1.34 (0.07) | -1.35 (0.07)
  Wakefulness/Alertness Score | -0.96 (0.06) | -1.00 (0.06)
  Energy Score | -1.28 (0.07) | -1.21 (0.07)
  Ability to Focus/Sustain Attention Score | -0.99 (0.06) | -1.02 (0.06)
  Ability to Remember/Recall Information Score | -0.91 (0.06) | -0.85 (0.06)
  Ability to Find Words Score | -0.69 (0.05) | -0.71 (0.05)
  Sharpness/Mental Acuity Score | -0.79 (0.05) | -0.85 (0.06)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.910, ANCOVA — This is the p-value for the Total Score; ANCOVA main effect F test
Statistical Analysis 2: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.882, ANCOVA — This is the p-value for the Motivation/Interest/Enthusiasm Score; ANCOVA main effect F test
Statistical Analysis 3: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.657, ANCOVA — This is the p-value for the Wakefulness/Alertness Score; ANCOVA main effect F test
Statistical Analysis 4: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.457, ANCOVA — This is the p-value for the Energy Score; ANCOVA main effect F test
Statistical Analysis 5: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.737, ANCOVA — This is the p-value for the Ability to Focus/Sustain Attention Score; ANCOVA main effect F test
Statistical Analysis 6: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.404, ANCOVA — This is the p-value for the Ability to Remember/Recall Information Score; ANCOVA main effect F test
Statistical Analysis 7: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.808, ANCOVA — This is the p-value for the Ability to Find Words Score; ANCOVA main effect F test
Statistical Analysis 8: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.431, ANCOVA — This is the p-value for the Sharpness/Mental Acuity Score; ANCOVA main effect F test

8. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total and Individual Scores at Week 8
Description: The SDS is a participant-rated assessment. Total scores range from 0-30 with higher values indicating greater disruption in the participant's work/social/family life. Items 1-3 assess the effect of the participant's symptoms on work/school schedule, social life/leisure activities, and family life/home responsibilities, respectively. Item scores are 0-10; higher values indicate greater disruption. Number of unproductive days and days lost in past week (symptom related) were reported. LS Mean Value was calculated from an ANCOVA model with terms of treatment, pooled investigator, and baseline.
Time Frame: Baseline, 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 211 | 209
units on a scale
  SDS Total Score | -7.55 (0.40) | -7.67 (0.41)
  SDS Work Score | -2.42 (0.14) | -2.29 (0.14)
  SDS Family Score (N=212, 210) | -2.51 (0.16) | -2.67 (0.16)
  SDS Social Score (N=212, 210) | -2.56 (0.16) | -2.72 (0.16)
  SDS Days Lost Score (N=208, 204) | -0.55 (0.11) | -0.60 (0.11)
  SDS Days Unproductive Score (N=209, 205) | -1.78 (0.13) | -1.89 (0.13)
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.821, ANCOVA — This is the p-value for the SDS Total Score; ANCOVA main effect F test
Statistical Analysis 2: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.491, ANCOVA — This is the p-value for the Item 1 (Work) Score; ANCOVA main effect F test
Statistical Analysis 3: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.451, ANCOVA — This is the p-value for the Item 2 (Family) Score; ANCOVA main effect F test
Statistical Analysis 4: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.443, ANCOVA — This is the p-value for the Item 3 (Social) Score; ANCOVA main effect F test
Statistical Analysis 5: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.719, ANCOVA — This is the p-value for the Item 4 (Days Lost) Score; ANCOVA main effect F test
Statistical Analysis 6: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.517, ANCOVA — This is the p-value for the Item 5 (Days Underproductive) Score; ANCOVA main effect F test

9. Secondary Outcome: Percentage of Participants Who Relapsed During 8 Weeks
Description: Relapse is defined as achieving a Montgomery-Asberg Depression Rating Scale (MADRS) total score≥16 at any time after baseline. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline through 8 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline result.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 243 | 237
percentage of participants | 11.9 | 11.0
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.776, Fisher Exact

10. Secondary Outcome: Number of Days From Baseline to Relapse as Defined by Montgomery-Asberg Depression Rating Scale (MADRS) Total Score ≥16 During 8 Weeks
Description: The number of days from baseline to the first relapse is defined as reaching a MADRS Total Score≥16. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Censored participants were included in the Kaplan-Meier analysis, the minimum and maximum time to relapse have been calculated and reported here. Median time to relapse and quartiles could not be computationally calculated using the Kaplan-Meier procedure due to low event rate and high completion rate (censored).
Time Frame: Baseline through 8 weeks
Population: Number of participants in each treatment group having time to relapse plus the participants censored. Duloxetine had 200 participants censored and escitalopram had 199 participants censored.
Measure: Number; unit: days
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 229 | 225
days
  Minimum Number of Days from Baseline | 4.00 | 4.00
  Maximum Number of Days from Baseline | 81.00 | 68.00
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; The log-rank test was conducted using Kaplan-Meier Product-Limit method; Test type: Superiority or Other; p = 0.691, Log Rank

11. Secondary Outcome: Percentage of Participants Who Discontinue Due to Lack of Efficacy During 8 Weeks
Description: Percentage of participants who discontinue after baseline due to lack of efficacy in the investigator's opinion.
Time Frame: Baseline through 8 weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Escitalopram
Number analyzed (Participants) | 244 | 239
percentage of participants | 2.0 | 1.3
Statistical Analysis 1: Comparison: Duloxetine vs Escitalopram; Test type: Superiority or Other; p = 0.724, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Duloxetine | Escitalopram
Serious Adverse Events (participants affected / at risk) | 3/244 | 3/239
Other Adverse Events (participants affected / at risk) | 130/244 | 100/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=244) | Escitalopram (N=239)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=244) | Escitalopram (N=239)
Constipation (Gastrointestinal disorders) | 23 (23) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 13 (14) | 8 (8)
Nausea (Gastrointestinal disorders) | 26 (26) | 28 (28)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Dizziness (Nervous system disorders) | 7 (8) | 15 (15)
Headache (Nervous system disorders) | 16 (16) | 20 (20)
Somnolence (Nervous system disorders) | 14 (15) | 8 (9)
Anxiety (Psychiatric disorders) | 9 (9) | 1 (1)
Insomnia (Psychiatric disorders) | 17 (21) | 10 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days